CLINICAL TRIAL: NCT02816502
Title: Hippocampal Plasticity of Young Adults With Childhood Adversity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mclean Hospital (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Diane Yan, Assistant Neuroscientist, Mclean Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016P000335
Record Dates: First submitted 2016-06-16; First posted 2016-06-28 (Estimated); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Depression; Anxiety
Keywords: childhood; adversity
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stress Management Skill Building Program A (Experimental): An eight week skill building group in which subjects meet with the teacher and other students in the group once a week, and complete homework and practice log during the week.
  Interventions: Behavioral: Stress Management Skill Building Program A
- Stress Management Skill Building Program B (Active Comparator): An eight week skill building group in which subjects meet with the teacher and other students in the group once a week, and complete homework and practice log during the week.
  Interventions: Behavioral: Stress Management Skill Building Program B

INTERVENTIONS:
Behavioral: Stress Management Skill Building Program A — Subject will meet with the instructor and other students in the group once a week and complete homework and track amount of practice during the week.
  Arms: Stress Management Skill Building Program A
Behavioral: Stress Management Skill Building Program B — Subject will meet with the instructor and other students in the group once a week and complete homework and track amount of practice during the week.
  Arms: Stress Management Skill Building Program B

SUMMARY:
This study investigates the clinical and neural effects of stress management skill building programs for young adults with childhood adversity. The investigators will recruit a total of 60 young adults (21-35 years old) who will be randomized into two different stress management skill building programs, both of which are 8 weeks long. MRI and psychological assessments will be acquired from all subjects before and after the intervention programs in order to investigate changes in clinical symptoms (such as depression, anxiety and stress) and hippocampus structure and function as well as other neural changes.

ELIGIBILITY:
Inclusion Criteria:

* having childhood adversity
* no history of psychiatric disorders of psychotic features or neurological disorders
* verified age between 21-35 years old;
* no suicidal attempts during the past six months;
* being determined by the clinician to have the capability to comply with the program requirements and not detrimental to other participants in the group;
* passing MRI eligibility criteria.
* provided written informed consent to participate in this study;
* committed to meeting the requirement of refraining from using marijuana or illicit drugs.

Exclusion Criteria:

* psychosis
* active suicidal attempts during the past 6 months
* psychoactive substance abuse
* MRI exclusion criteria

Ages: 21 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2020-07-07 (Actual)

PRIMARY OUTCOMES:
Changes in hippocampal subfield gray matter density measured with high resolution structural MRI at 3T | before and after the 8-week intervention

SECONDARY OUTCOMES:
Changes in stress level measured by the Perceived Stress Scale (PSS) | before and after the 8-week intervention
Changes in severity of depression symptom measured by Beck Depression Inventory (BDI) | before and after the 8-week intervention
Changes in severity of anxiety symptom measured by State-Trait Anxiety Inventory (STAI) | before and after the 8-week intervention

CONTACTS AND LOCATIONS:
Overall Officials: Diane Joss, PhD, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States